CLINICAL TRIAL: NCT02728882
Title: Single Arm, Two Phase, Multicenter Clinical Trial to Evaluating the Efficacy and Safety of the CAR-T for Recurrent or Refractory Diffuse Large B Cell Lymphoma
Brief Title: Study Evaluating the Efficacy and Safety With CAR-T for Recurrent or Refractory Diffuse Large B Cell Lymphoma
Acronym: EECBL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sinobioway Cell Therapy Co., Ltd. (Industry)
Collaborators: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACCO-2015-06-02
Record Dates: First submitted 2016-03-29; First posted 2016-04-05 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Lymphoma
Keywords: Lymphoma CAR-T
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): Name:The Chimeric Antigen Receptor T Cell Immunotherapy (CAR-T) Dosage form：injection Dosage:100ml/time Frequency:0 days，the first day,the fourth day,the seventh day,28 days,31 days,34 days.
  Duration:Total seven times.
  Interventions: Biological: CD19-targeted CAR-T cells

INTERVENTIONS:
Biological: CD19-targeted CAR-T cells — This study have only one arm that is CAR-T experimental arm. Firstly all participators will be attended the screening, who passed the screening for the treatment of CAR-T cells, the CAR-CD19-modified T cells can recognize and kill tumor cells in the body，follow-up 35 months.

SUMMARY:
This single-arm, multicenter Phase 2 study will treat the patients who have Recurrent or refractory diffuse large B cell lymphoma with an infusion of the patient's own T cells that have been genetically modified to express a chimeric antigen receptor (CAR) that will bind to tumour cells that express the EPCAM protein on the cell surface.The study will determine if these modified T cells help the body's immune system eliminate tumour cells.The trial will also study the safety of treatment with CAR-T,how long CAR-T cells stay in the patient's body and the impact of this treatment on survival.

DETAILED DESCRIPTION:
This is a single-arm, multicenter Phase 2 study to evaluate the efficacy and safety of the CAR-T for Recurrent or refractory diffuse large B cell lymphoma.The study will be conducted using a phase I/II design. The study will have the following sequential phases: Part A (screening leukapheresis,cell product preparation, and cytoreductive chemotherapy) and Part B (treatment and follow-up). The follow-up period for each participant is approximately 35 months after the final CAR-T infusion. The total duration of the study is expected to be approximately 3 years. A total of 24 patients may be enrolled over a period of 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed by pathological biopsy in patients with diffuse large B cell lymphoma by standard solution treatment is invalid or recurrence of refractory, and by flow cytometry or pathological immunohistochemical examination, confirmed the tumor cell surface expression positive intervention molecular targets, mainly for the CD19 (+) and/or CD20 (+).
2. Age 3 to 75 years old, both male and female;
3. Is expected to survive more than 3 months;
4. Physical condition is good: 0-2 score ECOG score;
5. In group of four weeks before Canon imaging examination evaluation body tumor load, recommend line PET - CT examination.
6. General requirements peripheral blood as basic, normal blood T lymphocytes in peripheral blood count must >= 0.2 x10^9 / L;
7. No obvious abnormal heart, liver, kidney, no large wounds that haven't healed on the body;
8. Into groups to participate in voluntarily, good adherence, can cooperate test observation, childbearing age women must be 7 days before starting treatment expert pregnancy test and the results were negative, and signed a written informed consent form.

Exclusion Criteria:

1. The recurrent or refractory patients with diffuse large B cell lymphoma.
2. Organ failure, such as heart: Class III and IV; liver: to Child grading of liver function grade C; kidney: kidney failure and uremia stage; lung: symptoms of severe respiratory failure; brain: disorder of consciousness;
3. Existing serious acute infection, uncontrollable, or have fester sex and chronic infection, wound in delay no more;
4. Patients with significant graft versus host disease (GVHD) after organ transplant history or allogeneic hematopoietic stem cell transplantation;
5. Systemic autoimmune diseases or immunodeficiency disease, patients with allergic constitution;
6. Coagulation abnormalities and severe thrombosis;
7. Pregnancy and lactation women;
8. Any other chronic disease patients who have been treated with immune agents or hormone therapy;
9. Patients who have participated in other clinical trials or other clinical trials in the past 30 days;
10. The Investigator believe the patients should not participate in this experiment.

Ages: 3 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-07-02 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Objective Reaction Rates | 0 to 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Kangsheng Gu, PI, Principal Investigator — Chief physician
Locations (1):
- The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No
No plans to share data.

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338